CLINICAL TRIAL: NCT02706288
Title: The Effects of a Calorie Restricted, Very Low Fat Plant-based Diet and Multi-component Exercise Program on Metabolic Health in Metabolically Abnormal Obese Adults
Brief Title: Effects of a Calorie Restricted, Very Low Fat Plant-based Diet and Multi-component Exercise Program on Metabolic Health
Acronym: PE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201512088
Record Dates: First submitted 2016-02-16; First posted 2016-03-11 (Estimated); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Obesity; Insulin Resistance
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weight loss with diet with exercise (Experimental): Persons with obesity with blood glucose concentrations higher than recommended and a moderate to high amount of fat in the liver (people with metabolically abnormal obesity) will be tested before and after ~7-10% weight loss. Following baseline testing, participants will be placed on a caloric-restricted plant-based very-low-fat (PB) diet and an exercise program until ~7-10% weight loss is achieved; they will then be re-tested so that pre- and post-intervention outcomes can be compared.
  Interventions: Other: Weight loss with very low fat plant-based diet and regular exercise

INTERVENTIONS:
Other: Weight loss with very low fat plant-based diet and regular exercise — Participants will lose ~7-10% of their body weight while on a calorie-restricted very low fat plant-based (PB) diet and performing exercise 6 days/week (4 sessions/week under direct supervision). The macronutrient composition of the diet is approximately 70% of energy from carbohydrate, 15% from protein, and 15% from fat. Food will be provided in the form of take-out meals and will be picked up by participants during weekly study visits with a weight management dietitian. To promote adherence to the diet and exercise intervention, subjects will participate in a lifestyle intervention program that includes dietary and behavioral education topics. Treatment will be provided in weekly individual or group sessions depending on subject availability. (Note: this is the only intervention for the study; the hyperinsulinemic euglycemic clamp is not an intervention but is the gold standard for evaluating insulin sensitivity, a primary study outcome.)

SUMMARY:
The purpose of this study is to understand how weight loss by a very low fat plant-based diet with an exercise program affects metabolic and cardiovascular health in overweight adults at high risk for disease. Outcome measures will include assessment of insulin sensitivity, β-cell function, body fat distribution, skeletal muscle and adipose tissue biology, cardiovascular function, cardiorespiratory fitness, muscular strength, immune function, and the gut microbiome.

DETAILED DESCRIPTION:
Reduced energy intake and increased physical activity have profound effects on cardiometabolic health as assessed by insulin sensitivity, β-cell function, serum lipids, intra-abdominal fat mass, intrahepatic triglyceride content, and blood pressure, and is the cornerstone of treatment for people with obesity. However, the specific additional therapeutic effects of regular exercise in conjunction with diet-induced weight loss are not clear. In addition, the optimal dietary macronutrient composition needed to reduce cardiometabolic risk is not known. The use of a very low fat, plant-forward diet is becoming increasingly popular to treat people with obesity and is the only diet therapy that is reimbursed by Medicare in the treatment of people with coronary heart disease.

Participants will undergo nutritional counseling and have supervised exercise training 4 days per week plus unsupervised exercise sessions performed 2 days per week until 7-10% weight loss is achieved. Meals will be provided and food diaries will be kept during weight loss. Tests before and after the intervention will include muscular strength and aerobic fitness, cardiovascular assessments, glucose tolerance tests, hyperinsulinemic euglycemic clamp test for insulin sensitivity, muscle biopsies, body composition scans, blood tests, and urine and stool collections.

The overarching goal of this project is to conduct a comprehensive characterization of weight loss induced by using a PB diet with regular exercise in people with obesity, prediabetes and insulin resistance, followed by a comparison of the effects of this study with those from another study that is evaluating the effect of the same amount of weight loss induced by using a PB diet alone, without exercise. Specifically, we will evaluate changes in body composition, body fat distribution, cardiopulmonary function, muscle strength, the plasma proteome, insulin sensitivity, beta-cell function, systemic inflammation, muscle cellular metabolic pathways, and the gut microbiome to determine cellular, multiorgan, and whole-body effects of PB diet alone and PB diet plus exercise. Accordingly, this study will fill two important gaps in our knowledge that have considerable physiological and clinical significance; the data from this study will provide: 1) a better understanding of the effects of calorie restriction-induced weight loss plus exercise on a series of key outcome measures, and 2) the potential additional benefit of adding regular exercise to a plant-forward diet.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤55 years
* BMI ≥30.0 and ≤50.0 kg/m²
* HbA1c ≥5.7%, or fasting plasma glucose concentration ≥100 mg/dl, or 2-hr OGTT plasma glucose concentration ≥140 mg/dl

Exclusion Criteria:

* Medical, surgical, or biological menopause
* Previous bariatric surgery
* Structured exercise >2 days/week for ≥35 minutes of intense exercise (e.g., jogging, activity that causes heavy breathing and sweating) or ≥150 min per week of structured exercise (e.g., brisk walking)
* Unstable weight (>4% change during the last 2 months before entering the study)
* Significant organ system dysfunction (e.g., diabetes requiring medications, severe pulmonary, kidney or cardiovascular disease)
* Cancer or cancer that has been in remission for <5 years
* Polycystic ovary syndrome
* Major psychiatric illness
* Conditions that render subject unable to complete all testing procedures (e.g., severe ambulatory impairments, limb amputations, or metal implants that interfere with imaging procedures; coagulation disorders)
* Use of medications that are known to affect the study outcome measures (e.g., steroids, non-statin lipid lowering medications) or increase the risk of study procedures (e.g., anticoagulants) and that cannot be temporarily discontinued for this study
* Use of antibiotics in last 60 days
* Smoke cigarettes, use marijuana >2 x/week, or use of illegal drugs
* Men who consume >21 units (e.g. glass of wine or bottle of beer) of alcohol per week and women who consume >14 units of alcohol per week
* Pregnant or lactating women
* Vegans, vegetarians, those with lactose intolerance and/or severe aversions/sensitivities to eggs, fish, nuts, wheat and soy, and/or any individuals with food allergies that induce an anaphylactic response
* Persons who are not able to grant voluntary informed consent
* Persons who are unable or unwilling to follow the study protocol or who, for any reason, the research team considers not an appropriate candidate for this study, including non-compliance with screening appointments or study visits

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity | An average of 4 months from baseline testing to 7-10% weight loss
  Liver and skeletal muscle insulin sensitivity will be assessed by hyperinsulinemic euglycemic clamp technique, before and after weight loss.

SECONDARY OUTCOMES:
Change in aerobic fitness | An average of 4 months from baseline testing to 7-10% weight loss
  Maximal oxygen consumption will be assessed using indirect calorimetry during a graded exercise test to volitional fatigue, before and after weight loss.
Change in muscular strength | An average of 4 months from baseline testing to 7-10% weight loss
  Muscle strength will be evaluated as the maximal amount of weight the participant is able to lift for one repetition (1 RM) for the following exercises: leg press, seated row, knee flexion, and chest press, before and after weight loss.
Change in fat mass and fat free mass | An average of 4 months from baseline testing to 7-10% weight loss
  Fat mass and fat free mass will be assessed using dual-energy x-ray absorptiometry (DXA) before and after weight loss.
Change in intra-hepatic triglyceride content | An average of 4 months from baseline testing to 7-10% weight loss
  Intra-hepatic triglyceride content will be assessed by magnetic resonance imaging (MRI) before and after weight loss.
Change in fasting plasma glucose | An average of 4 months from baseline testing to 7-10% weight loss
  Fasting plasma glucose concentrations will be evaluated from a fasting blood sample before and after weight loss.
Change in glycosylated hemoglobin (HbA1c) | An average of 4 months from baseline testing to 7-10% weight loss
  HbA1c will be evaluated from a fasting blood sample before and after weight loss.
Change in 24 hour glucose concentrations with feeding | An average of 4 months from baseline testing to 7-10% weight loss
  Glucose concentrations will be evaluated from frequent blood samples over a 24 h period, before and after weight loss, with the participant consuming mixed meals throughout the day.
Change in 24 hour metabolite concentrations with feeding | An average of 4 months from baseline testing to 7-10% weight loss
  Metabolite concentrations will be evaluated from frequent blood samples over a 24 h period, before and after weight loss, with the participant consuming mixed meals throughout the day.
Change in 24 hour hormone concentrations with feeding | An average of 4 months from baseline testing to 7-10% weight loss
  Hormone concentrations will be evaluated from frequent blood samples over a 24 h period, before and after weight loss, with the participant consuming mixed meals throughout the day.
Change in markers of inflammation | An average of 4 months from baseline testing to 7-10% weight loss
  Markers of inflammation will be evaluated from blood samples collected before and after weight loss.
Change in plasma proteome | An average of 4 months from baseline testing to 7-10% weight loss
  Plasma proteome will be evaluated from blood samples collected before and after weight loss.
Changes in gene expression in skeletal muscle tissue | An average of 4 months from baseline testing to 7-10% weight loss
  Gene expression in thigh muscle tissue will be evaluated before and after weight loss.
Changes in body weight | An average of 4 months from baseline testing to 7-10% weight loss
  Body weight will be measured before and after weight loss.
Changes in body mass index | An average of 4 months from baseline testing to 7-10% weight loss
  Body mass index will be calculated from weight and height before and after weight loss.
Change in exosome-mediated intercellular signaling | An average of 4 months from baseline testing to 7-10% weight loss
  Signaling between cells and organs will be examined by isolating exosomes (small extracellular vesicles) from blood
Change in gut microbiome | An average of 4 months from baseline testing to 7-10% weight loss
  Gut microbiota, meta-transcriptome (bacterial RNA sequencing to determine what proteins can be made by the microbiota) and the meta-metabolome (metabolites made by the microbiota) will be assessed before and after weight loss.
Change in beta-cell function | An average of 4 months from baseline testing to 7-10% weight loss
  Beta-cell function will be assessed from a modified oral glucose tolerance test before and after weight loss.
Change in insulin clearance | An average of 4 months from baseline testing to 7-10% weight loss
  Beta-cell function will be assessed from a modified oral glucose tolerance test and during the 24-hour study performed before and after weight loss.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
All of the data from individual subjects will be maintained confidentially and their names and identities will not be disclosed in any published document.

REFERENCES:
- [Derived] Beals JW, Kayser BD, Smith GI, Schweitzer GG, Kirbach K, Kearney ML, Yoshino J, Rahman G, Knight R, Patterson BW, Klein S. Dietary weight loss-induced improvements in metabolic function are enhanced by exercise in people with obesity and prediabetes. Nat Metab. 2023 Jul;5(7):1221-1235. doi: 10.1038/s42255-023-00829-4. Epub 2023 Jun 26. PMID 37365374